CLINICAL TRIAL: NCT00392119
Title: The Clinical Evaluation of the Stereotactic, MR Guided, Laser Interstitial Thermal Therapy (LITT ) for the "Minimal Invasive" Treatment of Brain Metastasis and Primary Brain Tumors - a Phase I Study With Direct Patient Benefice
Brief Title: MR Guided Laser Interstitial Thermal Therapy for the "Minimal Invasive" Treatment of Brain Metastasis and Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioTex, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUROLITT
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Brain Neoplasms; Brain Tumor; Brain Cancer; Recurrent Brain Tumor
Keywords: MR-guided therapy; Laser interstitial thermal therapy; brain metastasis; Magnetic Resonance Thermal imaging (MRTI)
MeSH Terms: conditions — Brain Neoplasms

INTERVENTIONS:
Device: MR-guided Laser Interstitial Thermal Therapy System

SUMMARY:
The purpose of this study is to determine if the stereotactic, MR guided, laser interstitial thermal therapy treatment technique can be safety and efficiently used for human brain metastasis and primary brain tumors.

DETAILED DESCRIPTION:
This new "minimally invasive" technique has been tested so far, with success, on animal brain tumor models and on human liver metastasis.

The main purpose of this study is to determine if the stereotactic, MR guided, laser interstitial thermal therapy treatment technique can be safety and efficiently used for the human brain metastasis and primary brain tumors.

As secondary objectives for this clinical study, the following are to be explored:

* Eventual evaluation of the eventual mid and long term post-intervention complications,
* Evaluate the contra indication for the technique,
* Evaluate and optimize clinical and logistic intervention protocols,
* Evaluate the mean duration for the procedure,
* Evaluate the mean cost for the procedure

The clinical trial will include a statistical sample of 12-18 treatments and will run over a period of 18 months. The inclusion period will be for 6 months and the patients will be followed up during 12 months post intervention.

The clinical trial will be performed at the Lariboisiere University Hospital of Paris and the patients will be coming from all the Assistance Publique de Paris ( APHP ) hospitals

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with brain metastasis located in the brain hemispheres
* Patient with a brain metastasis smaller or equal to 4 cm in diameter
* Patient with primary brain tumor smaller or equal to 4 cm in diameter
* Patient previously treated with other therapeutic techniques ( radio-therapy, chemotherapy, immunotherapy) which have failed.

Exclusion Criteria:

* Patients less than 18 years old,
* Patients presenting contra indication for MRI studies
* Patient for which the primary cancer is melanoma or kidney tumors
* Patients having a mean life duration longer than 3 months (due to the primary cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-10; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
12 month morbidity and mortality

SECONDARY OUTCOMES:
Mid and long term post-intervention complications,
Contra indication for the technique,
Optimize clinical and logistic intervention protocols,
Mean procedure duration
Mean procedure cost

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Carpentier, M.D./ Ph.D., Principal Investigator — Hospital Lariboisiere, Paris, France; Eric Vicaut, Ph.D., Study Chair — Hospital Lariboisiere, Paris, France; Daniel Reizine, M.D., Study Director — Hospital Lariboisiere, Paris, France
Locations (1):
- Hospital Lariboisiere, Paris, France

REFERENCES:
- [Derived] Carpentier A, McNichols RJ, Stafford RJ, Guichard JP, Reizine D, Delaloge S, Vicaut E, Payen D, Gowda A, George B. Laser thermal therapy: real-time MRI-guided and computer-controlled procedures for metastatic brain tumors. Lasers Surg Med. 2011 Dec;43(10):943-50. doi: 10.1002/lsm.21138. Epub 2011 Nov 22. PMID 22109661